CLINICAL TRIAL: NCT04886895
Title: Motor Training Intervention for Infants at High-Risk for Cerebral Palsy: Feasibility and Acceptability
Brief Title: Motor Training for Infants With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Karen Harpster, Associate Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0305
Record Dates: First submitted 2021-04-29; First posted 2021-05-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
Keywords: motor skills; occupational therapy; physical therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Single cohort
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Infants randomized to the usual care arm will receive usual care for 4 months. Therapy services provided to infants at this age vary in terms of frequency, location, and provider. Usual care is prescribed by the child's primary care provider (PCP), and in this population, usual care typically consists of one or both of the following: Early intervention therapy services provided by the state or Therapy in an outpatient clinic. Control group participants will be offered the Let's Move interventions after 16 weeks of control group.
  Interventions: Other: Let's Move Motor Intervention
- Intervention group: Let's Move (Experimental): Infants randomized to the Let's Move intervention group will be scheduled for therapy one time per week for 16 sessions (approximately 30-60 minutes per session). The intervention setting will involve both in-person (CCHMC clinic or in-home) and telehealth (in-home, video-based) sessions. The therapist will provide the caregivers with home programs to complete between therapy sessions (5 days per week). The home program will be based on the infant's goals set collaboratively between the caregiver and the evaluating therapist at the baseline assessment using the Canadian Occupational Performance Measure (COPM). At least half of the intervention sessions will be video recorded to assess feasibility and monitor intervention fidelity.
  Interventions: Other: Let's Move Motor Intervention

INTERVENTIONS:
Other: Let's Move Motor Intervention — Let's Move intervention will be administered and videotaped with infant/caregiver dyads. Therapy will occur weekly (30-60 minutes per session) for 16 weeks, alternating between clinic and home (video telehealth) sessions. Each month, we will attempt to schedule two clinic-based sessions followed by 2 telehealth-based sessions

SUMMARY:
The intervention in this study, Let's Move, is a motor intervention for infants at risk for cerebral palsy. We will test the feasibility and acceptability of the intervention as well as preliminary effectiveness.

DETAILED DESCRIPTION:
The aims of this study are to test the feasibility, acceptability, and operationalize a novel motor intervention, called "Let's Move" delivered using a combined clinic and home (video telehealth) therapy model.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment: between 3-8 months corrected age
* Caregivers fluent in English
* Preterm infants with objectively defined severe diffuse white matter abnormality on MRI at term OR
* High-risk infants (e.g., preterm, neonatal hypoxic-ischemic encephalopathy, perinatal stroke) with moderate-severe injury on structural MRI or cranial ultrasound (e.g., basal ganglia/thalamic signal intensity, cystic periventricular leukomalacia, encephalomalacia, large stroke, and/or severe intraventricular/periventricular hemorrhage) at around term-equivalent age or before Neonatal Intensive Care Unit discharge AND either:

  * "Absent" fidgety movements based on the Prechtl General Movement Assessment (GMA) between 3-4 months corrected age OR
  * A score of 56 or below on the Hammersmith Infant Neuromotor Examination (HINE) between 3-6 months corrected age (31)

Exclusion Criteria:

* Medical conditions that restrict active participation such as oxygen dependence
* Infants with significant visual deficits defined by the inability to track an object horizontally
* Living in a remote location prohibiting drives to the hospital every other week.

Ages: 3 Months to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change on Peabody Developmental Scales - Second Edition before and after intervention and follow-up | Baseline,16 weeks, 28 weeks
  Motor test

SECONDARY OUTCOMES:
Change on Pediatric Evaluation of Disability Inventory-Computer Adaptive Test before and after intervention and follow-up | Baseline,16 weeks, 28 weeks
  Parent reported test for functional performance
Change on Canadian Occupational Performance Measure before and after intervention and follow-up | Baseline,16 weeks, 28 weeks
  Caregivers perception of child's performance on functional goals
Change on Hammersmith Infant Neurological Exam before and after intervention and follow-up | Baseline,16 weeks, 28 weeks
  Neurological exam
Preverbal visual assessment (PreViAs | Enrollment, 4 months later, 8 months later
  Screening tool for the development of visual maturation

CONTACTS AND LOCATIONS:
Overall Officials: Karen Harpster, PhD, OTR/L, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided